CLINICAL TRIAL: NCT06643299
Title: PURE-LC - Probiotic Use for Recovery Enhancement From Long COVID
Brief Title: Probiotic Use for Recovery Enhancement From Long COVID-19
Acronym: PURE-LC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Gottlieb, Professor of Emergency Medicine, Vice Chair of Research, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 24082903
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Long COVID; Post-Acute Sequelae of COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic Arm (Active Comparator): Probiotic pill taken once daily
  Interventions: Drug: Probiotic Agent
- Placebo Arm (Placebo Comparator): Identical placebo pill taken once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Probiotic Agent — BlueBiology: Ultimate Care probiotic pill taken once daily for a four-month period.
  Other Names: BlueBiotics: Ultimate Care
  Arms: Probiotic Arm
Other: Placebo — Placebo produced to be identical in taste and appearance to the probiotic agent, taken once daily for a four-month period.
  Arms: Placebo Arm

SUMMARY:
The goal of this clinical trial is to learn if probiotics can improve symptoms and quality of life in participants with Long COVID.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if probiotics can improve symptoms and quality of life in participants with Long COVID. The main questions it aims to answer are:

1. Do probiotics reduce the number and severity of symptoms in those with Long COVID?
2. Do probiotics improve the physical and mental health quality of life in those with Long COVID?
3. Do probiotics improve return to work and daily activities in those with Long COVID?

Researchers will compare probiotics to a placebo (a look-alike substance that contains no probiotics) to see if probiotics work to treat Long COVID.

Participants will take the study medication (placebo or probiotic) for 4 months. They will then cross over (take the other medication) for an additional 4 months. Participants will complete a survey at baseline, 4 months, and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years who report Long COVID with persistent symptoms at the time of study initiation

Exclusion Criteria:

* No longer have symptoms consistent with LC
* Are unable to take the study medication daily
* Are currently pregnant or planning to become pregnant over the course of the study
* Are currently breastfeeding
* Have been diagnosed with an immune-compromising condition
* Are currently taking immunosuppressants
* Do not speak English as a primary language
* Are regularly taking probiotics
* Are enrolled in another Long COVID study with an intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in Long COVID Severity | Baseline, Four, and Eight Months
  Defined as the percentage change from moderate-to-severe Long COVID to mild Long COVID using the Long COVID Symptoms and Severity Score (LC-SSS) tool between groups with subgroup analysis by Long COVID trajectory

SECONDARY OUTCOMES:
Difference in LC-SSS Total Score | Baseline, Four, and Eight Months
  Defined as the change in the LC-SSS total score between groups with subgroup analysis by individual symptom scores and Long COVID trajectory
Difference in Quality of Life | Baseline, Four, and Eight Months
  Defined as the change in score for PROMIS-29 physical and mental health and the PROMIS SF-Cognitive Function 8a scale between groups with subgroup analysis by Long COVID trajectory
Difference in Return to Work and Activity | Baseline, Four, and Eight Months
  Defined as the change in the Work Productivity and Activity Impairment tool scores between groups with subgroup analysis by Long COVID trajectory

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No